CLINICAL TRIAL: NCT03775655
Title: Low Dose Hyperbaric Bupivacaine and Dexmedetomidine as an Adjuvant, Caesarean Section: Randomized Controlled Trial
Brief Title: Low Dose Hyperbaric Bupivacaine and Dexmedetomidine as an Adjuvant, Caesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Ashraf Nasr, Assisstant Lecturer Anesthesia, Intensive care and Pain management - Faculty of Medicie - Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9076411
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cesarean Section; Spinal Anesthesia; Dexmedetomidine
Keywords: Cesarean Section; Intrathecal Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LD-DEX (Active Comparator): This group will receive 7mg hyperbaric bupivacaine (about 1.4 ml of hyperbaric bupivacaine 0.5%) and 10μg dexmedetomidine (10 unit by U-100 insulin syringe using a preservative free dexmedetomidine 100μg/ml).
  Interventions: Drug: Dexmedetomidine
- Control group (No Intervention): This group will receive 12 mg hyperbaric bupivacaine (about 2.2 ml of hyperbaric bupivacaine 0.5%).

INTERVENTIONS:
Drug: Dexmedetomidine — 10μg dexmedetomidine will be added to the injectate to be injected intrathecally
  Other Names: Precedex
  Arms: LD-DEX

SUMMARY:
The aim of this study is to evaluate the effectiveness of low dose scheme with dexmedetomidine as an adjuvant. Taking in consideration optimum intraoperative surgical conditions, best post-operative pain free experience, and more stable hemodynamic.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnant women
* Singleton gestation
* American Society of Anaesthesiologists (ASA) physical status classes II and I

Exclusion Criteria:

* Preterm pregnancy (<37 wks. gestation)
* Multiple gestation
* Cardiovascular disease (e.g., preeclampsia, hypertension) and the use of antihypertensive medications
* Asthma and allergy to non-steroidal anti-inflammatory drugs
* Conditions that prevent spinal anaesthesia
* Failed spinal block and conversion to general anaesthesia
* A history of established chronic pain
* Drug addiction
* A psychiatric disorder
* Inability to communicate effectively

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Density of motor and sensory blockade | Intraoperative
Haemodynamic stability and total doses of IV fluids and vasopressors | Intraoperative
Time to first postoperative rescue analgesic request | 24 hour

SECONDARY OUTCOMES:
The intraoperative patient and surgeon satisfaction (successful delivery) | Intraoperative
The peak sensory level of block | Intraoperative
Time from intrathecal injection to peak sensory block level | Intraoperative
The time to two sensory block segment regression | Intraoperative and 24 hour
Degree and duration of motor block | Intraoperative and 24 hour
Intraoperative analgesic supplementation during operation | Intraoperative
Postoperative pain scores for 24 hours | 24 hour
Frequency and total dose of postoperative analgesics | 24 hour
Intraoperative and postoperative sedation scores | Intraoperative and 24 hour
Incidence of side effects: nausea, vomiting, shivering, pruritus, respiratory depression, and desaturation. | Intraoperative and 24 hour
Hospital in stay | 24 hour
Time to S1 level sensory regression | Intraoperative and 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mamdoh Lotfy, Prof. Dr., Study Chair — Faculty of Medicine - Menoufia University; Safaa M Helal, Prof. Dr., Study Chair — Faculty of Medicine - Menoufia University; Wesameldin A Soltan, Dr., Study Director — Faculty of Medicine - Menoufia University
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt